CLINICAL TRIAL: NCT00565123
Title: A Single- Centre, Randomised Study Of The Clinical And Microbiological Efficacy Of Decreasing The Dosage Of Levofloxacin 0,5% Eye Drops As Compared To Standard Eye Drop Dosage In Patients With Bacterial Conjunctivitis
Brief Title: Study of Efficacy of Levofloxacin 0.5% Ophthalmic Solution Administered Three Times a Day for Bacterial Conjunctivitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laser Microsurgery Centre, Poland (Other)
Collaborators: Katedra I Klinika Okulistyki II Wydz. Lek. AM w Warszawie, (Unknown); University Hospital No 1 Wroclaw (Other); MedSource Polska (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LF- 12/2003
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Bacterial Conjunctivitis
Keywords: bacterial conjunctivitis levofloxacin fluoroquinolone
MeSH Terms: conditions — Conjunctivitis, Bacterial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Experimental dosage
  Interventions: Drug: 0.5% levofloxacin eye drops
- Group B (Active Comparator): Classical dosage
  Interventions: Drug: 0.5% levofloxacin eye drops

INTERVENTIONS:
Drug: 0.5% levofloxacin eye drops — 0.5% levofloxacin eye drops three times daily to each eye for 5 days
  Arms: Group A
Drug: 0.5% levofloxacin eye drops — 0.5% levofloxacin eye drops 2 hours on days 1 and 2, and then every 4 hours on days 3-5 (up to 4 times per day)
  Arms: Group B

SUMMARY:
The aim of the study is to evaluate the clinical and microbiological efficacies of three times daily administration of levofloxacin 0,5% eye drops as compared to the more frequent dosing (up to 8 times a day during the first 2 days and up to 4 times a day during the next 3 days) in patients with bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 70 years of age
* Patients with Conjunctivitis (defined as the presence of three cardinal signs: conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection)
* Patients who have given and signed informed consent
* The ability and willingness to comply with all study procedures

Exclusion Criteria:

* Insulin Dependent Diabetes Mellitus (IDDM)
* Patients with keratitis or hordeolum
* Glaucoma
* Sjogren's Syndrom and "Sick Eye's Syndrom".
* Ectropion, entropion;
* Using contact lenses during the study
* Poor visual acuity in the other eye
* Prior and concurrent concomitant treatment glycocorticosteroids, immunosupressive therapy, if these treatments have not stopped at least 3 months prior to the start of the study;
* Concurrent use of non- steriodal anti- inflammatory drugs (NSAIDs), with the exception of low- dose aspirin. (see par. 11.5)
* Prior and concurrent systemic antibiotic treatment during last 7 days before the beginning the study.(see par. 11.5)
* Concurrent other eye drops
* All ocular surgeries which were performed less than 6 months before the beginning of the study.
* Any clinical condition, which, in the opinion of the investigator would not allow safe completion of the protocol.
* History of any malignancy within the past 5 years prior to study entry, except basal cell or squamous cell skin carcinoma.
* Hypersensitivity to fluoroquinolons and benzalkonium chloride;
* Intended or ascertained pregnancy or lactation;
* Participation in a clinical trial within last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the clinical cure. | 7(+-1) days

SECONDARY OUTCOMES:
The secondary efficacy end point was the microbiological eradication. | 7(+-1) days

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Szaflik, MD,Ph.D., Principal Investigator — Laser Microsurgery Centre; Department of Ophthalmology, Medical University of Warsaw
Locations (1):
- Centrum Mikrochirurgii Oka Laser, Warsaw, Masovian Voivodeship, Poland